CLINICAL TRIAL: NCT04859244
Title: First-in-Human Evaluation of the Safety, Tolerability, and Pharmacokinetics of Orally Administered GS-441524 in a Healthy Human Volunteer
Brief Title: First-in-Human Study of Orally Administered GS-441524 for COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Copycat Sciences LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CC-2021-001
Record Dates: First submitted 2021-04-19; First posted 2021-04-26 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-04

CONDITIONS: COVID-19
Keywords: GS-441524; remdesivir; GS-5734; Copycat Sciences; Gilead Sciences; COVID-19; antiviral
MeSH Terms: conditions — COVID-19 | interventions — GS-441524

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part 1: GS-441524 (QD, 7 days) (Experimental): 750 mg GS-441524 administered QD for 7 days
  Interventions: Drug: GS-441524
- Part 2: GS-441524 (TID, 3 days) (Experimental): 750 mg GS-441524 administered TID for 3 days
  Interventions: Drug: GS-441524

INTERVENTIONS:
Drug: GS-441524 — 750 mg administered as a solution
  Other Names: Parent nucleoside of remdesivir

SUMMARY:
This is a two-part study is to evaluate the multi-day safety, tolerability, and pharmacokinetics (PK) of orally administered GS-441524 in a healthy human volunteer.

DETAILED DESCRIPTION:
Part 1: 750 mg GS-441524 administered once daily (QD) for 7 days. Part 2: 750 mg GS-441524 administered three times daily (TID) for 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Negative pregnancy test at screening and prior to dosing
* Minimum body weight of 50 kg and body mass index (BMI) of 18-32 kg/m2

Exclusion Criteria:

* Use of other investigational drugs within 28 days of dosing
* Positive pregnancy test
* Abuse of alcohol or drugs
* Other clinically significant medical conditions or laboratory abnormalities

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Emergence of treatment-related adverse events (AEs) | Day 7
  Treatment-related AEs are defined as significant changes to blood chemistry (CBC, CMP) or 6-lead ECG.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Parameter: AUC0-24h of GS-441524 in Parts 1 and 2. | Intensive PK: Day 1 to Day 7
  AUC0-24h is defined as the concentration of drug over time between time 0 to time 24 hours.
PK Parameter: AUClast of GS-441524 in Parts 1 and 2. | Intensive PK: Day 1 to Day 7
  AUClast is defined as the concentration of drug from time zero to the last observable concentration.
PK Parameter: T1/2 of GS-441524 in Parts 1 and 2. | Intensive PK: Day 1 to Day 7
  T/2 is defined as the estimate of the terminal elimination half-life of the drug
PK Parameter: Cmax of GS-441524 in Parts 1 and 2. | Intensive PK: Day 1 to Day 7
  Cmax is defined as the maximum observed concentration of drug.
PK Parameter: Tmax of GS-441524 in Parts 1 and 2. | Intensive PK: Day 1 to Day 7
  Tmax is defined as the time (observed time point) of Cmax.
PK Parameter: Clast of GS-441524 in Parts 1 and 2. | Intensive PK: Day 1 to Day 7
  Clast is defined as the last observable concentration of drug.
PK Parameter: Tlast of GS-441524 in Parts 1 and 2. | Intensive PK: Day 1 to Day 7
  Tlast is defined as the time (observed time point) of Clast.
PK Parameter: AUCtau of GS-441524 in Parts 1 and 2. | Intensive PK: Day 1 to Day 7
  AUCtau is defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval).

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Yan, Principal Investigator — Copycat Sciences
Locations (1):
- Copycat Sciences Study Site, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 6 months after publication
Access Criteria: Materials available upon request

REFERENCES:
- [Background] Humeniuk R, Mathias A, Cao H, Osinusi A, Shen G, Chng E, Ling J, Vu A, German P. Safety, Tolerability, and Pharmacokinetics of Remdesivir, An Antiviral for Treatment of COVID-19, in Healthy Subjects. Clin Transl Sci. 2020 Sep;13(5):896-906. doi: 10.1111/cts.12840. Epub 2020 Aug 5. PMID 32589775
- [Background] Tempestilli M, Caputi P, Avataneo V, Notari S, Forini O, Scorzolini L, Marchioni L, Ascoli Bartoli T, Castilletti C, Lalle E, Capobianchi MR, Nicastri E, D'Avolio A, Ippolito G, Agrati C; COVID 19 INMI Study Group. Pharmacokinetics of remdesivir and GS-441524 in two critically ill patients who recovered from COVID-19. J Antimicrob Chemother. 2020 Oct 1;75(10):2977-2980. doi: 10.1093/jac/dkaa239. PMID 32607555
- [Background] Davis MR, Pham CU, Cies JJ. Remdesivir and GS-441524 plasma concentrations in patients with end-stage renal disease on haemodialysis. J Antimicrob Chemother. 2021 Feb 11;76(3):822-825. doi: 10.1093/jac/dkaa472. No abstract available. PMID 33152758
- [Background] Yan VC, Muller FL. Advantages of the Parent Nucleoside GS-441524 over Remdesivir for Covid-19 Treatment. ACS Med Chem Lett. 2020 Jun 23;11(7):1361-1366. doi: 10.1021/acsmedchemlett.0c00316. eCollection 2020 Jul 9. PMID 32665809
- See also: Preliminary results — https://osf.io/am5s8/
- Available data/document: Individual Participant Data Set — https://osf.io/am5s8/ — Supplementary Table 1: Blood chemistry (CBC, CMP) results. Supplementary Table 2: Plasma concentrations of GS-441524 at indicated timepoints.